CLINICAL TRIAL: NCT05546554
Title: Randomized Placebo-Controlled Crossover Trial of Suvorexant for Sleep in Children With Autism
Brief Title: Trial of Suvorexant for Sleep in Children With Autism
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Antonio Hardan, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB-67222; 1P50HD109861 (NIH)
Record Dates: First submitted 2022-09-12; First posted 2022-09-21 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: Suvorexant; Sleep; clinical trial; autism
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suvorexant, then Placebo (Experimental): Participants will first receive Suvorexant for a 4-week period. A starting dose will be 5 mg at bedtime and can be increased by 5 mg only if needed and if well tolerated on a weekly basis until the maximum dose of 20 mg/day is reached. Participants will be maintained on the lowest effective dose.
  Participants will then receive Placebo (fake tablet) for a 4-week period. A starting dose will be 5 mg at bedtime and can be increased by 5 mg only if needed and if well tolerated on a weekly basis until the maximum dose of 20 mg/day is reached. Participants will be maintained on the lowest effective dose.
  Interventions: Drug: Suvorexant; Drug: Placebo
- Placebo, then Suvorexant (Experimental): Participants will first receive Placebo (fake tablet) for a 4-week period. A starting dose will be 5 mg at bedtime and can be increased by 5 mg only if needed and if well tolerated on a weekly basis until the maximum dose of 20 mg/day is reached. Participants will be maintained on the lowest effective dose.
  Participants will then receive Suvorexant for a 4-week period. A starting dose will be 5 mg at bedtime and can be increased by 5 mg only if needed and if well tolerated on a weekly basis until the maximum dose of 20 mg/day is reached. Participants will be maintained on the lowest effective dose.
  Interventions: Drug: Suvorexant; Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant — 5 mg (and up to 20 mg) Suvorexant given orally
  Other Names: Belsomra
Drug: Placebo — Matching Placebo given orally

SUMMARY:
The purpose of this study is to examine the effect of suvorexant on sleep in children and adolescents with Autism Spectrum Disorder (ASD). Suvorexant is a selective, dual orexin receptor antagonist (DORA) used for the treatment of sleep onset difficulties and/or sleep maintenance. To accomplish this, the investigators will use a randomized double-blind placebo-controlled crossover 8-week study design to examine the effect of suvorexant on sleep physiology as assessed by polysomnography (PSG), actigraphy, circadian rhythm, and clinical measures.

ELIGIBILITY:
Inclusion criteria:

Participants will meet the following

* Outpatients between 13 and 17 years of age at time of consent
* Diagnostic and Statistical Manual, 5th edition (DSM-5) criteria for Autism Spectrum Disorder (ASD) on the basis of clinical evaluation, confirmed with the Autism Diagnostic Interview-Revised (ADI-R) and the Autism Diagnostic Observation Schedule, 2nd Ed (ADOS-2)
* Males and females
* Availability of polysomnography (PSG) and/or actigraphy data
* Sleep disturbances as assessed using Children's Sleep Habits Questionnaire (CSHQ) with a score of 41 or higher and sleep efficiency of 85% or less and/or total sleep time less than 7 hours and/or wake after sleep onset of more than 30 minutes as measured by polysomnography (PSG) or actigraphy
* care provider who can reliably bring participant to clinic visits, provide trustworthy ratings, and interacts with participant on a regular basis
* stable medications for at least 2 weeks, with the exception of Prozac which is required to be stable for at least 4 weeks
* no planned changes in psychosocial and biomedical interventions during the trial
* willingness to provide additional saliva samples and participate in key study procedures (i.e., safety measurements every visit, PSG at weeks 4 and 8, and wear the actigraphy watch for 2 weeks before the beginning of trial as well as during the 8 weeks of the trial).
* requirement of dual protection contraception use in females who are sexually active and are of childbearing potential. Dual use contraceptive methods involve the use of both a hormonal method (oral contraceptives, long-acting reversible contraceptives, etc.) and a barrier method (condoms).

Exclusion criteria:

Participants will be excluded if one or more of the following is met

* active suicidal ideation or DSM-5 diagnosis of severe depression, substance use disorder, schizophrenia, schizoaffective disorder, or psychotic disorder
* unstable medical problems: migraine, asthma, seizure disorder, significant physical illness (e.g., anaphylaxis, serious liver, renal, or cardiac pathology), obstructive sleep apnea and severe hepatic insufficiency
* evidence of a metabolic, or infectious etiology for the participant's autism on the basis of medical history, neurologic history, and available tests for inborn errors of metabolism
* pregnant or sexually active females not using a reliable method of contraception (urinary tests for pregnancy will be employed in this study)
* individuals taking beta-blockers (local or systemic), benzodiazepines, antiepileptic medications, melatonin and antihistamines
* history of hypersensitivity to suvorexant
* history of severe side effects from suvorexant
* history of adequate trial of suvorexant
* current use of any medications known to interact with suvorexant such as medications inhibiting CYP3A
* history of narcolepsy

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in sleep architecture as measured by polysomnography (PSG), examples include sleep latency and non-rapid eye movement (NREM) | Baseline, Week 4 and Week 8

SECONDARY OUTCOMES:
Change from baseline in sleep efficiency as measured by actigraphy | Baseline, Week 4 and Week 8

OTHER OUTCOMES:
Change from baseline on Children's Sleep Habits Questionnaire (CSHQ) subscale scores | Baseline, Week 4 and Week 8
Change from baseline on Aberrant Behavior Checklist, Second Edition (ABC-2) subscale scores | Baseline, Week 4 and Week 8
Change from baseline on Parent Sleep Habits Questionnaire Parent (PSHQ) scores | Baseline, Week 4 and Week 8
Change from baseline on Clinical Global Impression Scale (CGI) scores | Baseline, Week 4 and Week 8
Change from baseline on Child Behavior Checklist (CBCL) scores | Baseline, Week 4 and Week 8
Change from baseline on Social Responsiveness Scale, Second Edition (SRS-2) scores | Baseline, Week 4 and Week 8
Change from baseline on Repetitive Behavior Scale - Revised (RBS-R) scores | Baseline, Week 4 and Week 8
Change from baseline on Sensory Profile Questionnaire (SPQ) scores | Baseline, Week 4 and Week 8
Change from baseline on Stanford Social Dimension Scale (SSDS) scores | Baseline, Week 4 and Week 8
Change from baseline on Dimensional Assessment of Repetitive Behaviors (DARB) score | Baseline, Week 4 and Week 8
Change from baseline on NEuroPSYchological Assessment, 2nd Edition (NEPSY-2) Affect Recognition scores | Baseline, Week 4 and Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Y. Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will submit de-identified clinical data to the NIMH Data Archive (NDA) data repository.
URL: https://nda.nih.gov/nda/data-contribution.html